CLINICAL TRIAL: NCT05067504
Title: Prospective, Evaluator-blind, Multicenter Study to Assess the Safety and Effectiveness of Treatment With the Octave System for Lifting the Eyebrow and Improving the Appearance of the Face and Neck
Brief Title: Effectiveness and Safety of the Octave System for Lifting the Eyebrow and Improving the Appearance of the Face and Neck
Acronym: LIFT-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M960101001
Record Dates: First submitted 2021-09-22; First posted 2021-10-05 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Eyebrow Lift; Improved Appearance of the Face and Neck

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will receive a single Octave-Ultherapy treatment of the brow, face, and neck.
Masking Description: While there was only one arm, Outcome Assessors were masked to pre- vs post-treatment images.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Octave-Ultherapy treatment (Experimental): Octave-Ultherapy treatment of the brow, face, and neck.
  Interventions: Device: Octave-Ultherapy treatment

INTERVENTIONS:
Device: Octave-Ultherapy treatment — Micro-focussed ultrasound delivered below the surface of the skin.

SUMMARY:
This study was conducted to evaluate the effectiveness and safety of the Octave System to lift the eyebrow and improve the appearance of the face and neck.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate eyebrow/upper-face laxity.
* Mild to moderate fine lines, wrinkles, and laxity of the face and neck.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Scarring in area(s) to be treated.
* Active implants (e.g., pacemakers or defibrillators), ports, or metallic implants in area(s) to be treated.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (3):
- United States (2):
  - Merz Investigational Site #0010358, Vista, California
  - Merz Investigational Site #0010101, Coral Gables, Florida
- Merz Investigational Site #0010436, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigational sites in the United States.
Pre-assignment Details: Of the 65 screened subjects, 15 subjects exited as screen failures and 50 subjects (10 subjects in Stage 1 and 40 subjects in Stage 2) were enrolled to receive a single Octave-Ultherapy treatment of the brow, face, and neck in this study.
Groups:
- Stage 1: Octave-Ultherapy Treatment: Subjects received a single Octave-Ultherapy treatment of the brow, face, and neck on Day 1 of Stage 1 with two transducers.
- Stage 2: Octave-Ultherapy Treatment: Subjects received a single Octave-Ultherapy treatment of the brow, face, and neck on Day 1 of Stage 2 with up to four transducers.
Period: Period 1 (Day 90)
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Started | 10 | 40
Completed | 10 | 40
Not Completed | 0 | 0
Period: Period 2 (Day 180)
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Started | 10 | 40
Completed | 6 | 39
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not reconsented for Period 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety population (SP) included all subjects who were enrolled and treated with the Octave System.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment | Total
Number analyzed (Participants) | 10 | 40 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (9.65) | 51.0 (8.42) | 50.5 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 36 | 44
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 25 | 28
  Not Hispanic or Latino | 7 | 15 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 35 | 41
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treated Subjects With Eyebrow Lift at Day 90
Description: Improvement in eyebrow lift was determined by three evaluators after comparing Day 90 photographs with baseline photographs. Lift was concluded if at least two evaluators reported "eyebrow lift" in the Day 90 photographs as compared to baseline.
Time Frame: Day 90
Population: Intent-to-treat (ITT) population included all subjects who were enrolled.
Measure: Number; unit: percentage of subjects
Groups:
- Stage 2: Octave-Ultherapy Treatment": Subjects received a single Octave-Ultherapy treatment of the brow, face, and neck on Day 1 of Stage 2 with up to four transducers.
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment"
Number analyzed (Participants) | 10 | 40
percentage of subjects | 80.0 | 67.5

2. Secondary Outcome: Percentage of Treated Subjects With Eyebrow Lift at Day 180
Description: Improvement in eyebrow lift was determined by three evaluators after comparing Day 180 photographs with baseline photographs. Lift was concluded if at least two evaluators reported "eyebrow lift" in the Day 180 photographs as compared to baseline.
Time Frame: Day 180
Population: ITT. Here "overall number of subjects analyzed" were subjects who were eligible for this outcome measure. The results for this outcome measure across both stages were estimated using the ITT population with multiple imputations.
Measure: Number; unit: percentage of subjects
Groups:
- Stage 1: Octave-Ultherapy Treatment": Subjects received a single Octave-Ultherapy treatment of the brow, face, and neck on Day 1 of Stage 1 with two transducers.
Arm/Group | Stage 1: Octave-Ultherapy Treatment" | Stage 2: Octave-Ultherapy Treatment"
Number analyzed (Participants) | 7 | 40
percentage of subjects | 81.7 | 64.7

3. Secondary Outcome: Percentage of Treated Subjects With Eyebrow Lift of at Least 0.5 Millimeter (mm) at Day 90 and Day 180
Description: Eyebrow lift position on frontal view was measured by calculating the differences in eyebrow height. Standard images of the subject's face were collected before treatment, and at Day 90 and Day 180 to visualize and quantify changes in the treated regions.
Time Frame: Day 90 and Day 180
Population: ITT.
Measure: Number; unit: percentage of subjects
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Number analyzed (Participants) | 10 | 40
percentage of subjects
  Day 90 | 20.0 | 27.5
  Day 180 | 16.7 | 30.8

4. Secondary Outcome: Change From Baseline in FACE-Q Satisfaction With Forehead and Eyebrows Score (Rasch-transformed) at Day 90 and Day 180, as Assessed by Subject
Description: The FACE-Q is a set of standardized patient-reported outcome scales for subjects undergoing facial cosmetic procedures. The subject assessed satisfaction using the Face-Q Satisfaction with Forehead and Eyebrows module (1 [very dissatisfied] to 4 [very satisfied] scores; Rasch transformed score 0-100; higher scores meant better outcome).
Time Frame: At Baseline, Day 90 and Day 180
Population: ITT. Here, "number analyzed" signifies those subjects who were evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Number analyzed (Participants) | 10 | 40
score on a scale
  Day 90 | 10.1 (33.27) | 21.1 (22.12)
  Day 180: number analyzed (Participants) | 6 | 39
  Day 180 | 20.5 (11.48) | 22.7 (20.51)

5. Secondary Outcome: Change From Baseline in FACE-Q Satisfaction With Lower Face and Jawline Score (Rasch-transformed) at Day 90 and Day 180, as Assessed by Subject
Description: The FACE-Q is a set of standardized patient-reported outcome scales for subjects undergoing facial cosmetic procedures. The subject assessed satisfaction using the Face-Q Satisfaction with Lower Face and Jawline module (1 [very dissatisfied] to 4 [very satisfied] scores; Rasch transformed score 0-100; higher scores meant better outcome).
Time Frame: At Baseline, Day 90 and Day 180
Population: ITT. Here, "number analyzed" signifies those subjects who were evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Number analyzed (Participants) | 10 | 40
score on a scale
  Day 90 | 25.0 (27.22) | 28.9 (27.35)
  Day 180: number analyzed (Participants) | 6 | 39
  Day 180 | 37.2 (17.58) | 26.9 (28.66)

6. Secondary Outcome: Change From Baseline in FACE-Q Patient-Perceived Age Visual Analogue Scale (VAS) Rating at Day 90 and Day 180, as Assessed by the Subject
Description: For the FACE-Q Patient-perceived Age VAS, subjects were asked a question "How many years younger or older do you think you look compared with your actual age?". Perception of age compared to actual age, in years ranging from -15 years (best outcome) to +15 years (worst outcome).
Time Frame: At Baseline, Day 90 and Day 180
Population: ITT. Here, "number analyzed" signifies those subjects who were evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Number analyzed (Participants) | 10 | 40
score on a scale
  Day 90 | -0.9 (3.00) | -2.2 (3.55)
  Day 180: number analyzed (Participants) | 6 | 39
  Day 180 | -2.0 (3.16) | -2.4 (4.20)

7. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) Related to Octave-Ultherapy Treatment
Description: TEAEs were defined as adverse events (AEs) with onset or worsening on or after date of first administration of Octave-Ultherapy Treatment.
Time Frame: From first treatment on Day 1 up to the end of study on Day 180 (an average of 6 months)
Population: SP.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
Number analyzed (Participants) | 10 | 40
Participants | 4 | 6

ADVERSE EVENTS:
Time Frame: From first treatment on Day 1 up to the end of study on Day 180 (an average of 6 months)
Description: SP. The investigator reported AEs systematically at each visit.
Arm/Group | Stage 1: Octave-Ultherapy Treatment | Stage 2: Octave-Ultherapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/40
Other Adverse Events (participants affected / at risk) | 5/10 | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Octave-Ultherapy Treatment (N=10) | Stage 2: Octave-Ultherapy Treatment (N=40)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Octave-Ultherapy Treatment (N=10) | Stage 2: Octave-Ultherapy Treatment (N=40)
Application site pain (General disorders) | 2 | 2
Application site pruritus (General disorders) | 1 | 2
Application site urticaria (General disorders) | 1 | 2
Application site discomfort (General disorders) | 1 | 0
Application site dysaesthesia (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT05067504/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05067504/SAP_001.pdf